CLINICAL TRIAL: NCT01998100
Title: Maximizing Treatment Outcome in Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Mark B. Powers, Research Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS10-106
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Anxiety; Behavior Therapy; Prolonged Exposure; Exercise; Wellness; Post-traumatic; Stress
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prolonged Exposure + Exercise (Experimental)
  Interventions: Behavioral: Prolonged Exposure; Behavioral: Exercise
- Prolonged Exposure Alone (Active Comparator)
  Interventions: Behavioral: Prolonged Exposure

INTERVENTIONS:
Behavioral: Prolonged Exposure — 75-90 minute weekly psychotherapy sessions x 12 weeks, focused on gradually confronting distressing trauma-related memories and reminders.
Behavioral: Exercise — 30 minutes of moderate-intensity treadmill exercise prior to the Prolonged Exposure
  Arms: Prolonged Exposure + Exercise

SUMMARY:
The purpose of this study is to examine the efficacy of exercise + therapy to therapy alone to determine if they can improve the effects of prolonged exposure therapy (PE) in reducing symptoms of anxiety associated with Post-traumatic Stress Disorder (PTSD). In addition the two strategies (i.e., exercise + therapy and therapy alone condition) will be compared in terms of levels of brain-derived neurotrophic factor (BDNF). BDNF is a protein that helps to support the survival of existing neurons and stimulate the growth of new neurons and synapses. BDNF is important to learning and memory in general and therefore may be associated with the learning and memory as it relates to PE and corresponding symptoms PTSD improvement.

ELIGIBILITY:
Inclusion Criteria:

* You have PTSD.
* You are between the ages of 18 and 65.
* You have written physician approval/medical clearance to participate in an exercise protocol.
* You are currently taking no psychotropic medications or are able and willing to discontinue these medications prior to the first PE session.

Exclusion Criteria:

* You are currently participating in a structured exercise program.
* You have severe depression.
* You have any history of bipolar disorder, psychotic disorder, or obsessive compulsive disorder.
* You have a diagnosis of eating disorder, or substance abuse or dependence (excluding nicotine) within the past six months.
* You have any history of a suicide attempt, or are at a significant risk or self-harm or harm to others.
* You have ever been diagnosed with organic brain syndrome, mental retardation, or other cognitive dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
PTSD Symptoms | 3 months
  Self-report measure that assesses PTSD symptoms. Will be assessed at each visit throughout the three month protocol.

SECONDARY OUTCOMES:
BDNF (by blood sample) | 3 months
  Small blood sample taken twice (at the beginning and end of the 3 month protocol).
General Mood and Anxiety Symptoms | 3 months
  Self-report measures that assesses mood and anxiety. Will be assessed at each visit throughout the 3 month protocol.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Texas at Austin, Austin, Texas
  - Southern Methodist University, Dallas, Texas

REFERENCES:
- [Result] Powers MB, Medina JL, Burns S, Kauffman BY, Monfils M, Asmundson GJ, Diamond A, McIntyre C, Smits JA. Exercise Augmentation of Exposure Therapy for PTSD: Rationale and Pilot Efficacy Data. Cogn Behav Ther. 2015;44(4):314-27. doi: 10.1080/16506073.2015.1012740. Epub 2015 Feb 23. PMID 25706090